CLINICAL TRIAL: NCT06042634
Title: An Evidence-based Online Psychoeducation for Family Caregivers of People With Dementia: A Feasibility Study
Brief Title: A Feasibility Study of Online Psychoeducation for Family Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chan Hoi Man Jackie, Doctoral Student, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: online psychoeducation
Record Dates: First submitted 2023-09-08; First posted 2023-09-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Dementia
Keywords: family caregivers; online; psychoeducation; self-efficacy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Parallel arm of 1:1 ratio
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor was blinded to group allocation of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online psychoeducation (Experimental): The online psychoeducation was presented virtually via Zoom videoconferencing for synchronous group meeting. It has two core components: didactic teaching and active participation. The didactic teaching provided information support about dementia caregiving which was delivered via Powerpoint presentations. The programme allowed: (1) hands-on skill training opportunities to rehearse caregiving skills through simulation and written assignments; (2) sharing of caregiving experiences and learning vicariously from other participants through group discussion; (3) reflection on own caregiving approach; and (4) addressing negative emotions through practicing relaxation technique. Participants went through six-weekly psychoeducation sessions in a small group of five to eight. Each psychoeducation session consisted of didactic teaching and active participation which lasted for 120 minutes. Participants went through discussion, simulation and was given home assignment weekly.
  Interventions: Behavioral: Online psychoeducation
- Face-to-face psychoeducation (Active Comparator): Face-to-face psychoeducation had the same content and flow of presentation as online psychoeducation. The only difference was the mode of delivery which was presented physically in the community center.
  Interventions: Behavioral: Face-to-face psychoeducation

INTERVENTIONS:
Behavioral: Online psychoeducation — Online psychoeducation aimed to enhance the knowledge and skill of family caregivers of people with dementia, who could not physically attend in-person class. Knowledge covering dementia caregiving including disease nature, communication skill, stress and coping, daily care, management of behavioral and psychological symptoms of dementia, and future planning. The intervention provided opportunities to practice through simulation and weekly home assignment. There was a total of 6 sessions and provided weekly. Each session lasted for 2 hours. Participants had discussion with peers and coached by a facilitator. Online psychoeducation wad delivered via Zoom videoconferencing.
  Arms: Online psychoeducation
Behavioral: Face-to-face psychoeducation — Face-to-face psychoeducation has the same content and flow of presentation as online psychoeducation.
  Arms: Face-to-face psychoeducation

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and acceptability of online psychoeducation in the family caregivers of people with dementia living in the community. The main objectives it aims to answer are:

1. Is online psychoeducation feasible and acceptable to family caregivers of people with dementia?
2. What is the preliminary effect of online psychoeducation on caregiving self-efficacy in family caregivers of people with dementia?

DETAILED DESCRIPTION:
This study employed a quasi-experimental pretest-posttest design to compare online psychoeducation with conventional face-to-face psychoeducation. This study also included a qualitative study as process evaluation to explore the participants' experiences with the online psychoeducation.

Caregivers of people with dementia were recruited from two sources: elderly community centers and Facebook. Printed flyers were physically displayed in the elderly community centers and advertisements were posted on Facebook. Interested participants approached the principal investigator through telephone and were screened for eligibility. Informed consent was collected physically at the elderly community centers or via Google Forms.

The feasibility study required 30 participants per arm to test the intervention before a future definitive trial. Therefore, with two groups in this study, the total sample size was set at 60.

Participants recruited from the elderly community centers were allocated to the face-to-face group, whilst participants recruited from Facebook were allocated to the online group. The rationale for having a non-randomized design was to prevent potential contamination occurring due to information sharing among the participants. Participants were informed of the group allocation at the time of recruitment.

The sociodemographic data and outcomes were collected by an research assistant. All participants were also asked to complete the satisfaction questionnaire at T1. Questions for the satisfaction questionnaire and caregiving self-efficacy questionnaire were read out to participants.

Quantitative data were analyzed using the IBM SPSS Statistics version 26.0. Descriptive statistics were used to summarize the demographic data and the feasibility outcomes including recruitment rate, attrition rates, completion rate of intervention, participants' satisfaction score and completion rate of instrument. Chi-square test for the categorical variables and independent T-test for the continuous variables were used to examine the homogeneity of the participants in the two intervention groups. Analysis of Covariance was performed to examine between group differences in Revised Scale of Caregiving Self-Efficacy (RSCSE) score, with the respective pretest score as covariate. Paired T-test was also performed to examine within group differences in RSCSE score. Effect size was measured by dividing the mean difference within the group by the pooled standard deviation and reported as Cohen's d value. The cut-off points of small, medium and large effect size were 0.2, 0.5 and 0.8 respectively. All analysis was considered significant at p≤ 0.05 (2-tailed).

The audio-recorded interviews were transcribed verbatim for qualitative content analysis. The transcripts were managed with the support of Nvivo 14 for systematic organization of the data. The authors read the transcripts multiple times to get familiar with the data. They then coded the data and developed initial themes independently. Critical discussion and revision on the themes and subthemes were carried out until a consensus was reached. The main themes and subthemes were refined and named collaboratively. Illustrative quotes were selected through critical discussion between authors. The first author translated the quotes to English while the other authors helped with verification and proofreading.

ELIGIBILITY:
Inclusion Criteria:

* cognitively competent (i.e. Mini Mental State Examination ≥23)
* taking care of a family member diagnosed with dementia of mild to moderate stage and required assistance in physical activities of daily living (ADL) (i.e. score ≥2 on the ADL scale
* at least 5 hours of caregiving per week in the past month
* had low caregiving self-efficacy (i.e. score ≤3 on the Caregiving Competence Scale

Exclusion Criteria:

* currently participating in any other psychosocial interventional program
* had psychiatric illnesses and had active treatment
* did not had access to the Internet on any type of electronic device such as smart phone or laptop.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Sociodemographic background | Baseline
  Caregiver: Age, gender, marital status, relationship with care recipient, caregiving experience, education level, level of confidence in caregiving; Care recipient: age, gender, duration of dementia since diagnose, level of assistance required in activity daily living, stage of dementia
Recruitment rate | Through study completion, an average of 6 months
  The proportion of eligible subjects and consented to join the study.
Attrition rate | Through study completion, an average of 6 months
  The proportion of consented subjects who dropped out of the study. The reasons for attrition such as refusal were recorded.
Completion rate | Through study completion, an average of 6 months
  The proportion of participants who attended at least 4 out of 6 sessions.
Class attendance | Through study completion, an average of 6 months
  The proportion of participants who attended the class in each session
Completion rate of study instrument | Through study completion, an average of 6 months
  The proportion of participants who completed the study instrument
Satisfaction of intervention | On completion of intervention at 6 weeks
  Participants rated on the content, format and appropriateness of intervention on a 5-point Likert scale. The higher total score represented greater satisfaction with the intervention
Experience of online psychoeducation | On completion of intervention at 6 weeks
  Individual semi-structured interviews were conducted to explore the experience of online psychoeducation.

SECONDARY OUTCOMES:
Caregiving self-efficacy | Baseline and on completion of intervention at 6 weeks
  Participants completed the Revised Scale of Caregiving Self-efficacy. There are 15 questions in total and participant rated on a scale of 0-100 on each question. The mean score of 15 questions will be presented and the higher the score represented the higher level of caregiving self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Man Chan, master, Principal Investigator — Nethersole School of Nursing, Chinese University of Hong Kong
Locations (1):
- Nethersole School of Nursing, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Upon request to the principal investigator, Jackie Chan Hoi Man via email: 1010155350@link.cuhk.edu.hk
Supporting Information: SAP, ICF, CSR
Time Frame: 2 years after completion of study and for 5 years